CLINICAL TRIAL: NCT00376350
Title: Dose-Response/Efficacy of Manipulation for Chronic LBP
Brief Title: Dose of Spinal Manipulation for Chronic Low Back Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Western States (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mitchell Haas, Associate Vice President of Research, University of Western States
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01AT001908 (NIH); U01AT001908 (NIH)
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Chronic; Manipulation; Chiropractic; Massage
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome | interventions — Manipulation, Spinal; Ultrasonic Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High dose manipulation (Experimental): High dose spinal manipulation + ultrasound
  Interventions: Procedure: Spinal Manipulation; Procedure: Pulsed Ultrasound
- Moderate dose manipulation (Experimental): Moderate dose manipulation + low dose massage + ultrasound
  Interventions: Procedure: Spinal Manipulation; Procedure: Light Massage; Procedure: Pulsed Ultrasound
- Low dose manipulation (Experimental): low dose spinal manipulation + moderate dose massage + ultrasound
  Interventions: Procedure: Spinal Manipulation; Procedure: Light Massage; Procedure: Pulsed Ultrasound
- High dose masssage (Other): high dose massage + ultrasound
  Interventions: Procedure: Light Massage; Procedure: Pulsed Ultrasound

INTERVENTIONS:
Procedure: Spinal Manipulation — 5 minutes high velocity, low amplitude lumbar thrust
  Arms: High dose manipulation; Low dose manipulation; Moderate dose manipulation
Procedure: Light Massage — light pressure massage of the low back.
  Arms: High dose masssage; Low dose manipulation; Moderate dose manipulation
Procedure: Pulsed Ultrasound — 5 minutes pulsed ultrasound

SUMMARY:
This study will determine the number of visits to a chiropractor for spinal manipulation, light massage, and ultrasound necessary for optimal relief of chronic low back pain. The study will also determine the effectiveness of spinal manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Current episode of low back pain
* mechanical origin
* Threshold low back pain level

Exclusion Criteria:

* Contraindications to spinal manipulation or massage
* Complicating conditions that could confound clinical outcome
* Prophylactic use of prescription medication
* Health-related litigation, claims, or disability compensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Modified Von Korff Pain Scale for low back pain | baseline 1&2, 6, 12, 18, 24, 39, 52 weeks
Modified Von Korff Disability Scale | baseline 1&2, 6, 12, 18, 24, 39, 52 weeks

SECONDARY OUTCOMES:
Pain days | baseline 1&2, 6, 12, 18, 24, 39, 52 weeks
Disability days | baseline 1&2, 6, 12, 18, 24, 39, 52 weeks
Low back pain unpleasantness | baseline 2, 6, 12, 18, 24, 39, 52 weeks
Fear avoidance beliefs | baseline 2, 6, 12, 18, 24, 39, 52 weeks
General health status/QoL | baseline 2; 12, 24, 39, 52 weeks
Patient satisfaction | 12 wk
Healthcare utilization | baseline 2; 6, 12, 18, 24, 39, 52 weeks
Objective measures | Baseline 2, 6 wk
Bias monitoring | baseline 1&2; 6, 12, 18, 24, 39, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Haas, DC, MA, Principal Investigator — University of Western States
Locations (1):
- Western States Chiropractic College, Portland, Oregon, United States

REFERENCES:
- [Background] Haas M, Groupp E, Kraemer DF. Dose-response for chiropractic care of chronic low back pain. Spine J. 2004 Sep-Oct;4(5):574-83. doi: 10.1016/j.spinee.2004.02.008. PMID 15363431
- [Result] Haas M, Vavrek D, Peterson D, Polissar N, Neradilek MB. Dose-response and efficacy of spinal manipulation for care of chronic low back pain: a randomized controlled trial. Spine J. 2014 Jul 1;14(7):1106-16. doi: 10.1016/j.spinee.2013.07.468. Epub 2013 Oct 16. PMID 24139233
- [Result] Haas M, Vavrek D, Neradilek MB, Polissar N. A path analysis of the effects of the doctor-patient encounter and expectancy in an open-label randomized trial of spinal manipulation for the care of low back pain. BMC Complement Altern Med. 2014 Jan 13;14:16. doi: 10.1186/1472-6882-14-16. PMID 24410959
- [Result] Vavrek D, Haas M, Neradilek MB, Polissar N. Prediction of pain outcomes in a randomized controlled trial of dose-response of spinal manipulation for the care of chronic low back pain. BMC Musculoskelet Disord. 2015 Aug 19;16:205. doi: 10.1186/s12891-015-0632-0. PMID 26286532
- [Result] Vavrek DA, Sharma R, Haas M. Cost analysis related to dose-response of spinal manipulative therapy for chronic low back pain: outcomes from a randomized controlled trial. J Manipulative Physiol Ther. 2014 Jun;37(5):300-11. doi: 10.1016/j.jmpt.2014.03.002. PMID 24928639